CLINICAL TRIAL: NCT06799988
Title: NUTFINFORCE: THE IMPACT OF DIGITALLY DELIVERED LIFESTYLE PERFORMANCE MEDICINE INTERVENTION ON DEFENSE PERFORMANCE IN FINLAND
Acronym: NutFinForce
Status: Not yet recruiting | Type: Observational
Sponsor: University of Helsinki (Other)
Collaborators: Metropolia University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Kristiina Patja, Professor, University of Helsinki
Other Study IDs: University of Helsinki 250123
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: No Condition
Keywords: Nutrition; Eating habits; Digital; Behavior change; Performance medicine
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Digitally Delivered Lifestyle Performance Medicine intervention — Participating is realized by downloading the application to their phone with the privacy statement for participation in the study must be read and accepted before use can begin. Application can be removed at any stage. Intervention protocol and implementation responsibility is in the University of Helsinki and digital coaching tools is provided by the Metabite Ltd. Digital tool in the intervention is Metabite (https://www.metabite.com/) with specified version designed with the Finnish Defense Force. All content within the application is based on scientific evidence and has been reviewed for relevance and applicability to the Finnish context by local healthcare professionals

SUMMARY:
Summaries are in Finnish for attendees are availabe and reviewed in ethical approcval process

DETAILED DESCRIPTION:
Abstract in English Background: Physical and cognitive demands on military service are ever-increasing in the Finnish Defense Forces. The University of Helsinki and Center for Military medicine are conducting a pioneering research initiative known as the NutFinForce study. This innovative project aims to evaluate the impact of a digital delivered lifestyle intervention on the defense performance of Finnish conscripts.

Objective and Scope: The primary objective of the study is to enhance the physical and cognitive performance through targeted nutritional and lifestyle digital intervention. Equally we will assess the feasibility, acceptability, and cost-effectiveness of personalized digital health coaching and support for adopting healthier dietary and lifestyle habits. The aim is to foster long-term health benefits for public health and to improve national defense capability that isa a cumulative outcome for optimizing health of reserve.

Methodology: The intervention leverages a sophisticated digital platform that offers personalized guidance and support to participants. Special attention is paid to target group needs and military service as an environment in intervention design. Platform is accessible before, during, and after military service, ensuring opportunities for longitudinal and sustainable engagement and support. A large-scale implementation includes two sequential brigades (N=5000). Data collection will be conducted through the digital application platform used in the intervention.

Expected Outcomes: Key outcomes will include improvements in nutrition and eating patterns and perceived physical performance as swell as perceived cognitive sharpness/performance as a variable for outcome. The study will evaluate the cost-effectiveness of the intervention, providing important data for future policy and practice within the Finnish Defense Forces and NATO ally military forces.

Implications for Military Policy and Public Health: The findings from the NutFinForce study will have significant implications for military policy and practice. By demonstrating the benefits of digital health interventions that positively influence daily lifestyle behavior choices, the research could inform the development of future nutritional and lifestyle programs within the military. Moreover, the study's insights may have broader public health implications, highlighting the potential of digital health platforms to promote healthier behaviors and improve population health.

ELIGIBILITY:
Inclusion Criteria:

* The participants for the intervention are recruited along with the invitation process of the Finnish Defense Forces in such a way that it does not interfere with the actual goal itself: attending the military service.

Attendance for the intervention, suspension of the intervention or not attending is not known by the Defense Forces and does not influence terms of service

Exclusion Criteria:

* Not attending the military service

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The conscription of the Finnish Defense Forces is carried out nationally at the location specified in the conscription letter. For many years already, the conscripts will have had a digital intervention available for developing their physical fitness and an invitation to a phone application
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Eating habits and patterns | 24 moths
  Group based analyses of eating contents will include averages and patterns e.g. Total Energy Intake, Fruit and Vegetables and Nutrient-Dense Foods Percentage of total Daily Energy Intake Energy-Dense Beverages like Sugar Sweetened Beverages (SSBs) and fruit juice Individual Food Groups and macronutrients Energy-Dense Nutrient-Poor (Ed-Np) Foods Diet Quality Score Rating

SECONDARY OUTCOMES:
Nutirion component analyses | 24 moths
  Proportion of vegetable and fiber intake among users pre and post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided
All data will be managed according to a Data Management Plan compiled at the start of the project and divided into four steps: Data Collection, Storage and Documentation, and Data Sharing. All steps of the Data Management Plan that is following the data management protocols of the University of Helsinki

REFERENCES:
- See also: Study will run under the Helsinki Planetary Health Hub, at the Medical Faculty — https://www.helsinki.fi/en/researchgroups/helsinki-planetary-health/projects
- See also: Related Info — https://www.helsinki.fi/en/researchgroups/helsinki-planetary-health/projects